CLINICAL TRIAL: NCT04127474
Title: Expression of Trefoil Factors 2 and 3 and Adrenomedullin in Unstimulated Saliva Samples of Chronic Periodontitis Subjects With and Without Coronary Heart Disease
Brief Title: Expression of Trefoil Factors and Adrenomedullin in Subjects With Chronic Periodontitis and Coronary Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor, PhD guide, Director of Post Graduate Studies, Meenakshi Ammal Dental College and Hospital
Other Study IDs: MADC/IRB-XXIX/2019/468
Record Dates: First submitted 2019-10-14; First posted 2019-10-15 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Coronary Heart Disease; Periodontal Diseases
Keywords: periodontitis; saliva; trefoil factor; adrenomedullin; Coronary heart disease
MeSH Terms: conditions — Coronary Disease; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: 25 Generalized chronic periodontitis subjects without coronary heart disease.
- Group II: 25 Generalized chronic periodontitis subjects diagnosed with coronary heart disease.
- Group III: 25 Periodontally healthy subjects diagnosed with coronary heart disease.

SUMMARY:
To assess the demographic variables, periodontal parameters and to determine the expression of Trefoil factors 2 and 3 and Adrenomedullin in unstimulated saliva samples of periodontally healthy subjects with coronary heart disease and generalised chronic periodontitis subjects with and without coronary heart disease.

DETAILED DESCRIPTION:
A total of 75 subjects will be recruited for the study based on the power of the study.

The selected subjects will be divided into 3 groups based on inclusion and exclusion criteria.

GROUP I:25Generalized chronic periodontitis subjects without coronary heart disease.

GROUP II: 25Generalized chronic periodontitis subjects diagnosed with coronary heart disease.

GROUP III: 25Periodontally healthy subjects diagnosed with coronary heart disease.

Demographic variables, periodontal parameters and biochemical parameters will be measured in all three groups

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to participate in the study.
2. Patients within the age group of 30-65 years.
3. Patients should have ≥ 20 remaining natural teeth.
4. For Group I

   • Systemically healthy, Generalized chronic periodontitis subjects with 30% or more sites with clinical attachment loss (CAL) ≥ 2mm, radiographic evidence of alveolar crestal bone loss ≥ 2mm from the cemento-enamel junction.
5. For Group II

   • Generalized chronic periodontitis subjects with 30% or more sites with clinical attachment loss (CAL) ≥ 2mm, radiographic evidence of alveolar crestal bone loss ≥ 2mm from the cemento-enamel junction along with coronary heart disease.
6. For Group III • Periodontally healthy subjects with Probing pocket depth (PD) less than 4mm, bleeding on probing (BOP) at ≤15% of tooth sites, no periodontal treatment (Scaling and root planing or periodontal surgery) within the previous 6 months and without evident clinical signs of gingival inflammation along with the presence of coronary heart disease.

Exclusion Criteria:

1. Subjects with systemic conditions such as type I and type II diabetes mellitus, respiratory diseases, renal disease, liver disease, rheumatoid arthritis, allergy, advanced malignancies and HIV infection will be excluded from the present investigation.
2. For Group I, subjects on drugs such as corticosteroids, antibiotics, within 6 months of investigation will be excluded.
3. Current smokers and individuals who quit smoking less than 6 months.
4. Patients who have undergone periodontal therapy within the previous 6 months.
5. Pregnant women (pregnancy may alter the oral flora)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants from 30 years to 65 years will be recruited for the study. Subjects would be categorized into the above mentioned three groups based on their medical status.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-12-20 (Estimated); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
Trefoil factors 2 and 3 and Adrenomedullin expression in Chronic periodontitis patients with and without coronary heart disease | 12 months
  Expression of Trefoil factors 2 and 3 and Adrenomedullin using Enzyme Linked Immunosorbent Assay

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Mahendra, MDS, PhD, Study Director — Meenakshi Ammal Dental College
Locations (1):
- Meenakshi Ammal Dental College, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaiyarit P, Chayasadom A, Wara-Aswapati N, Hormdee D, Sittisomwong S, Nakaresisoon S, Samson MH, Pitiphat W, Giraud AS. Trefoil factors in saliva and gingival tissues of patients with chronic periodontitis. J Periodontol. 2012 Sep;83(9):1129-38. doi: 10.1902/jop.2011.110431. Epub 2011 Dec 19. PMID 22181686
- [Background] Suchetha A, Garg A, Lakshmi P, Bhat D, Sapna N, Apoorva SM. Adrenomedullin, periodontitis, diabetes-unraveling the equivocal relationship: A clinicobiochemical cross-sectional study. Contemp Clin Dent. 2013 Oct;4(4):454-9. doi: 10.4103/0976-237X.123040. PMID 24403788